CLINICAL TRIAL: NCT03570294
Title: Evaluation of Oxidative and Antioxidative Status of Pregnant Women Suffering From Threatened Preterm Birth During Tocolytic Treatment With Atosiban
Brief Title: Oxidative Stress in Women Treated With Atosiban for Impending Preterm Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Polish Mother Memorial Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015/I/17-GW
Record Dates: First submitted 2018-06-15; First posted 2018-06-26 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2018-06

CONDITIONS: Premature Birth
MeSH Terms: conditions — Premature Birth | interventions — atosiban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atosiban (Other): Total oxidant status (TOS), total antioxidant status (TAS) and oxidative stress index (OSI) values as well as 3-nitrotyrosine, carbonyl and thiol groups levels weill be measure using ELISA test in serum and plasma of 64 pregnant women before and after 48 hours of continuous administration of Atosiban.
  Interventions: Drug: Atosiban

INTERVENTIONS:
Drug: Atosiban — The initial dose of Atosiban (Tractocile, Ferring Pharmaceuticals A/S, Copenhagen, Denmark) will be give as a single intravenous bolus dose (6.75 mg in 0.9 ml isotonic sodium chloride solution). This will be follow immediately by intravenous infusion of 300 μg/min of Atosiban in 5% glucose for 3 hours, and then 100 μg/min for up to 48 hours. Venous blood samples from a forearm vein will take before and after 48 hours of continuous administration tocolytic therapy with Atosiban.
  Other Names: Tractocile

SUMMARY:
Oxidative stress is recognized as a important factor in the pathogenesis premature birth. Preterm birth is defined as delivery before 37 completed weeks of gestation and it is the leading cause of neonatal morbidity and mortality. The investigators conducted this analysis to investigate the safety of administration of Atosiban - a reversible, competitive antagonist of the oxytocin receptor in the treatment of preterm labor and its impact on the level of oxidative stress after 48 hours of tocolytic treatment.

DETAILED DESCRIPTION:
Atosiban (1-(3-mercaptopropanoic acid)-2-(O-ethyl-D-tyrosine)-4-L-threonine-8-L-ornithine-oxytocin) is licensed for clinical use in women suffering from threatened premature birth and is widely used in clinical practice in Europe because of its low side effect profile. The impact of Atosiban on pregnancy outcomes in women has been investigated in recent years and the research has shown its ability to reduce intracytoplasmic calcium release and downregulate prostaglandin synthesis as oxytocin receptor antagonist. While a role of Atosiban in the modulation of myometrial contractility is well-described, its effect on many other functions is not so well known.

The serum and plasma samples take for the measurement of total oxidant status (TOS), total antioxidant status (TAS), level of 3-nitrotyrosine (3-NT), and carbonyl and thiol groups will be stored at -70°C in aliquots for subsequent biochemical analysis and processed within two months.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women between 24-35 weeks' gestation receiving prenatal care due to the risk of premature birth
* intact membranes
* evidence of premature labor (regular, painful and persistent uterine contractions; cervical changes)

Exclusion Criteria:

* acute fetal distress
* other conditions requiring immediate delivery (eclampsia and severe pre-eclampsia, placenta previa, abruptio placenta)
* vaginal bleeding,
* premature rupture of membranes
* chorioamnionitis,
* fetal congenital malformations,
* intrauterine growth restriction,
* the use of any tocolytic drugs during pregnancy before admission to the hospital
* circulatory system diseases (e.g. heart defects, hypertension),
* symptoms of infection
* other diseases that may increase oxidative stress

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 64 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2018-06-10 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Delay preterm delivery for 48 hours | 48 hours
  Delay preterm delivery for 48 hours, thus allowing administration of corticosteroids to induce surfactant production in fetal lungs and improve neonatal outcome

SECONDARY OUTCOMES:
Apgar score | At birth
  Apgar score
Weight | At birth
  Weight
Incidence of duration of hospitalization | Up to 28 days after birth
  Incidence of duration of hospitalization
Time to delivery measured from start of Atosiban administration | Up to 15 weeks from start of Atosiban administration
  Time to delivery measured from start of Atosiban administration

CONTACTS AND LOCATIONS:
Overall Officials: Mariusz Grzesiak, Ph.D. MD, Principal Investigator — Department of Obstetrics, Perinatology and Gynecology, Polish Mother's Memorial Hospital-Research Institute
Locations (1):
- Department of Obstetrics, Perinatology and Gynecology, Polish Mother's Memorial Hospital-Research Institute, Lodz, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Study protocol, statistical analysis plan, informed consent form, clinical study report

REFERENCES:
- [Derived] Grzesiak M, Gaj Z, Kocylowski R, Suliburska J, Oszukowski P, Horzelski W, von Kaisenberg C, Banach M. Oxidative Stress in Women Treated with Atosiban for Impending Preterm Birth. Oxid Med Cell Longev. 2018 Dec 2;2018:3919106. doi: 10.1155/2018/3919106. eCollection 2018. PMID 30622667